CLINICAL TRIAL: NCT07174388
Title: A Prospective Study to Generate Precision External Controls in Advanced or Metastatic Non Small Cell Lung Cancer Patients
Brief Title: A Study in Non-Small Cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: N-Power Medicine (Industry)
Responsible Party: Sponsor
Other Study IDs: NPM-004
Record Dates: First submitted 2025-09-12; First posted 2025-09-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; External Control Arm; Non-Interventional; N-Power Medicine; Registry; Prospective
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Optional submission of archived tissue when available. Should originate from a prior diagnostic biopsy or surgical resection. Provision of archived tissue is optional and not required for study eligibility, enrollment, or continued participation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Cohort 1: Patients starting first line pembrolizumab or pembrolizumab in combination with a platinum doublet
- Cohort 2: Patients with KRASG12D mutation starting first or later line of therapy
- Cohort 3: Patients planned to have second line docetaxel or docetaxel in combination with ramucirumab with tumor without alterations in KRAS, EGFR, ALK, or ROS1
- Cohort 4: Patients with PD-L1 > 50% treated with single agent immuno-oncology therapy (IO) or dual IO agents as first line treatment.
- Cohort 5: Patients with PD-L1 < 50% without alterations in KRAS, EGFR, ALK, or ROS1
- Cohort 6: Patients with documented KRAS G12C mutation
- Cohort 7: Patients with non-G12C and non-G12D KRAS mutations
- Cohort 8: Patients with EGFR mutations with prior treatment with osimertinib in combination with chemotherapy or lazertinib in combination with amivantamab
- Cohort 9: Patients initiating single agent docetaxel or docetaxel and ramucirumab as third line of therapy

SUMMARY:
A study to create control arms using current and future information in patients with lung cancer that has spread who have already received chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years of age at the time of informed consent 2. Pathologically confirmed NSCLC 3 .ECOG Performance of >1 and fit for further systemic therapy on a NCCN approved regimen (within 4 weeks prior or 14 days after starting second line therapy) 4. Life expectancy of more than 3 months 5. Able to understand and sign informed consent *see protocol for cohort specific inclusion criteria*

Exclusion Criteria:

1. Unable to provide informed consent
2. Actively on a clinical trial of an investigational agent
3. Non protocol compliant baseline imaging scan (modality/coverage) prior to index date in patients included after the second or third line therapy has been initiated *see protocol for cohort specific exclusion criteria* -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic NSCLC receiving first, second or third line NCCN recommended therapies
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2026-01-07 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Assess Objective Response Rate (ORR) by cohort in patients with metastatic NSCLC treated in second or third line with NCCN recommended therapies | September 2025-April 2029

SECONDARY OUTCOMES:
Assess Progression Free Survival (PFS), Overall Survival (OS), and Time to Next Treatment (TTNT) by cohort in patients with metastatic NSCLC initiating second or third line treatment with NCCN recommended therapies. | September 2025-April2029

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Pacific Cancer Care, Monterey, California
  - Bayhealth Medical Center, Kent Campus, Dover, Delaware
  - Bayhealth Medical Center- Sussex Campus, Milford, Delaware

IPD SHARING:
Plan to Share IPD: Undecided
undecided